CLINICAL TRIAL: NCT01130727
Title: Randomized Clinical Trial, Placebo Controlled, With Parallel Groups to Investigate Whether Green Tea or Cocoa Extracts Improves Endothelial Dysfunction in Patients With Diabetes Mellitus and Nephropathy and Hypertension
Brief Title: The Effect of Green Tea or Cocoa Extracts in Endothelial Dysfunction in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Jose Butori Lopes de Faria, Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTCOCOA-01
Record Dates: First submitted 2010-05-18; First posted 2010-05-26 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathy; Arterial Hypertension
Keywords: diabetes mellitus; diabetic nephropathy; hypertension; green tea; cocoa; polyphenol; nitric oxide
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Hypertension | interventions — Tea; Long-Term Synaptic Depression; Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- green tea extract (Active Comparator)
  Interventions: Other: green tea extract
- Cocoa extract rich in polyphenols (Active Comparator)
  Interventions: Other: cocoa extract rich in polyphenols
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- cocoa extract with low polyphenol (Placebo Comparator)
  Interventions: Other: low polyphenol cocoa extract

INTERVENTIONS:
Other: green tea extract — 1.21g of green tea extract (965 mg of flavonols)
  Other Names: Green tea extract, sunphenon 90DCF-T, Tayo, CO., LTD
  Arms: green tea extract
Other: cocoa extract rich in polyphenols — 2.14 g of cocoa extract rich in polyphenols equivalent to 965 mg of polyphenols
  Other Names: Acticoa cocoa extract NCE-PO803-W41, Barry Callebaut, Belgium
  Arms: Cocoa extract rich in polyphenols
Other: placebo — placebo
  Arms: placebo
Other: low polyphenol cocoa extract — placebo
  Other Names: placebo cocoa extract, Barry Callebaut, Belgium
  Arms: cocoa extract with low polyphenol

SUMMARY:
The purpose of this study is to determine whether green tea or cocoa extracts are effective in improve endothelial dysfunction in patients with diabetes mellitus and nephropathy and arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* Diabetic nephropathy
* Hypertension

Exclusion Criteria:

* GFR < 30 ml/min/1.73m2
* Serum K > 5.5 mEq/L
* Age < 18 y
* Pregnancy
* Breast feeding
* Cocoa or green tea intolerance
* Alcohol and drugs abuse
* Incapacity to understand the information related to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation (FMD) | up to 4 hours

SECONDARY OUTCOMES:
arterial blood pressure and cardiac rate | up to 4 hours
plasma levels of flavonols | up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jose b Lopes de Faria, M.D., Principal Investigator — Universidade Estadual de Campinas, Unicamp
Locations (1):
- University Hospital, Campinas, São Paulo, Brazil